CLINICAL TRIAL: NCT05124925
Title: An Open-label, Non-randomized, Biopsy-based Mechanistic Study on Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Ianalumab in Patients With Sjögren's Syndrome
Brief Title: Biopsy Based Study to Understand Mechanism of Action of Ianalumab in Salivary Glands and Explore Relationships With Clinical Assessments.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAY736A2103; 2023-508957-24-00 (Registry Identifier: EU CT NUMBER)
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Sjogren Syndrome
Keywords: Sjogren syndrome; VAY736; Ianalumab; dry eyes; dry mouth
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes; Xerostomia | interventions — ianalumab

STUDY DESIGN:
Intervention Model Description: This is an open label study (with no control arm) with a 5 weeks screening period, a 6-month treatment period and a follow up period of up to 2 years after the last dose The study consists of a first Run-in Phase that includes Screening and Baseline period of 35 days. After signing the Informed Consent, participants will be assessed as per inclusion/exclusion criteria. All study participants who successfully pass the screening will be considered eligible for the treatment period.
  All eligible participants will enter the 6 months treatment period and will have the two other biopsies taken at the end of treatment (6 months after the screening) and end of the study (EOS) after blood B cell recovery (from 5 months up to 2 years after the last dose).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Ianalumab 300 mg subcutaneous monthly
  Interventions: Biological: Ianalumab

INTERVENTIONS:
Biological: Ianalumab — Ianalumab VAY736 150mg/1ml Solution for injection

SUMMARY:
This study aims at elucidating the mechanism of action of ianalumab in salivary glands and explore relationships with clinical assessments

DETAILED DESCRIPTION:
This is an open-label, non-randomized, biopsy-based mechanistic study on pharmacokinetics, pharmacodynamics, safety and tolerability of ianalumab in patients with Sjögren's syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed
2. Male and female patients 18 years of age or older at Screening
3. Confirmed Sjögren's syndrome according to the 2016 ACR/EULAR classification criteria
4. Seropositive for anti-Ro/SSA antibodies
5. Screening ESSPRI score ≥ 5
6. Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Use of other investigational drugs within 5 half-lives of enrollment or within 30 days whichever is longer, or longer if required by local regulations
2. Presence of another autoimmune rheumatic disease that is active and constitutes the primary illness
3. Prior use of ianalumab
4. History of receiving:

   o Any B-cell depleting therapies, other than ianalumab (e.g., rituximab, other anti-CD20 mAb, anti-CD22 mAb, or anti-CD52 mAb) administered within 36 weeks prior to randomization, or as long as B cell count is less than the lower limit of normal or baseline value prior to receipt of B cell-depleting therapy (whichever is lower)
5. Current use of prednisone >10 mg/day [or equivalent other corticosteroid] or dose change within 2 weeks prior to dosing
6. Prior treatment with any of the following within 6 months of baseline

   1. CTLA4-Fc Ig (abatacept)
   2. Anti-TNF-α mAb
   3. Intravenous Ig
   4. Plasmapheresis
   5. i.v. or oral cyclophosphamide
   6. i.v. or oral cyclosporine A
   7. Patients taking either hydroxychloroquine more than 400 mg/day or methotrexate more than 25 mg weekly or leflunomide at not stable dose within 3 months prior to dosing.
   8. iscalimab (anti-CD40)
   9. belimumab (anti-BAFF mAb)
7. Active viral, bacterial or other infections
8. History of major organ, hematopoietic stem cell or bone marrow transplant
9. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes (e.g., mAb of IgG1 class) or to any of the constituents of the study drug formulation (sucrose, L-histidine hydrochloride/L-histidine, polysorbate 20)
10. Required regular use of medications known to cause dry mouth/eyes as a regular and major side effect, and which have not been on a stable dose for at least 30 days prior to Screening, or any anticipated change in the treatment regimen during the course of the study
11. Receipt of live/attenuated vaccine within a 4-week period prior to baseline
12. History of primary or secondary immunodeficiency, or a positive HIV (ELISA and Western blot) test result
13. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin, in situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
14. History of head and neck radiation therapy or of having received radioactive iodine
15. Any one of the following screening values of CBC laboratory values:

    * Hemoglobin levels below 8.0 g/dL;
    * Total leukocyte count less than 2,000/μL;
    * Platelets <50 x 109/L (if between 50 and 80, the PI should check that it is linked to Sjögren's syndrome and not to any other disease);
    * Absolute neutrophil count (ANC) <1.0 x 109/L (one re-test is allowed during the screening period)
16. Positive serology for hepatitis B surface antigen (HBsAg).

    Positive serology for hepatitis B core antibody (HBcAb), except if all 3 following criteria are met:
    * Hepatitis B (HBV) quantitative PCR for viral DNA is negative (i.e., <10 IU)
    * Prophylactic treatment (with tenofovir or entecavir) initiated latest on day 1 and continued until 12 months after last treatment
    * Hepatitis B monitoring is implemented: HBsAg (and HBV DNA) tested every 4 weeks during treatment and at least every 12 weeks after end of treatment for the entire duration of the follow-up. Antiviral prophylaxis must be implemented while on study and up to 12 months after end of study treatment.
17. Positive hepatitis C test result. Participants with a positive HCV antibody test should have HCV RNA levels measured. Participants with positive (detectable) HCV RNA should be excluded.
18. Evidence of active tuberculosis (TB) infection (after anti-TB treatment, patients with history of or latent TB may become eligible according to national guidelines)
19. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
20. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 6 months after stopping of investigational medication. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) total hysterectomy or tubal ligation at least six weeks before taking investigational drug. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening and confirmed as successful). For female patients in the study, the vasectomized male partner should be the sole partner for that patient
    * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking investigational drug.

    Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

    If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the informed consent form (ICF).
21. Known contraindication to SonoVue (sulphur hexafluoride microbubbles) ultrasound contrast agent
22. Participants not registered in the social security system
23. Participants within the exclusion period of a preceding study
24. Any surgical, medical (e.g. uncontrolled hypertension, heart failure or diabetes) psychiatric or additional physical condition that the investigator feels may jeopardize the patient in case of participation in this study
25. People deprived of their liberty by a judicial or administrative decision (Article L1121-6 of the French Public Health Code)
26. Screening Labial minor salivary gland (LMSG) biopsy lymphocyte focus score < 0.3/4 mm2 or B/B+T ratio in the gland < 0.2 (20%)
27. Use of topical ocular prescription medications (excluding artificial tears, gels, lubricants) that have not been on a stable dose for at least 90 days prior to treatment, or any anticipated change in the treatment regimen during the course of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Change in logarithm of salivary gland B/B+T cell ratio | Week 25
  Change from baseline in logarithm of salivary gland B/B+T cell ratio at Week 25 (EOT)

SECONDARY OUTCOMES:
Number of participants with Adverse Events | 6 months treatment plus 2 years of follow-up
  Occurrence of treatment emergent adverse events (both serious and non-serious) during the study and occurrence of treatment emergent abnormal vital signs, laboratory and ECG data.
Change from baseline in disease activity at salivary gland level by ultrasound imaging | 6 months treatment plus 2 years of follow-up
  Changes in salivary gland tissue (parenchymal abnormalities, vascularization, perfusion and stiffness) by multimodal salivary gland ultrasound (SGUS) after treatment with ianalumab
Incidence of ADA positive patients | 6 months treatment plus 2 years of follow-up
  Serum anti-ianalumab antibody (ADA assay) and incidence of ADA positive patients as a measure of immunogenicity (IG) of ianalumab
Change of salivary flow | 6 months treatment plus 2 years of follow-up
  Defined as change in stimulated and unstimulated salivary flow from baseline
Serum ianalumab concentrations PK parameters Tmax | 6 months treatment plus 2 years of follow-up
  To assess the pharmacokinetics (PK) of ianalumab
Serum ianalumab concentrations AUCinf | 6 months treatment plus 2 years of follow-up
  To assess pharmacokinetics (PK) of ianalumab
Serum ianalumab concentrations C-max | 6 months treatment plus 2 years of follow-up
  To assess pharmacokinetiks (PK) of ianalumab
Serum ianalumab concentrations PK parameters AUC from dosing to the time of the last measurable concentrations (AUClast) | 6 months treatment plus 2 years of follow-up
  To assess the pharmacokinetics (PK) of ianalumab
Serum ianalumab concentrations PK parameters half life (T1/2) | 6 months treatment plus 2 years of follow-up
  To assess the pharmacokinetics (PK) of ianalumab
Serum ianalumab concentrations PK parameters AUC calculated to the end of a dosing interval (tau) at steady state | 6 months treatment plus 2 years of follow-up
  To assess the pharmacokinetics (PK) of ianalumab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com